CLINICAL TRIAL: NCT01277991
Title: Phase 1, Open-label, Randomized, Single-dose, 2-treatment, 2-period, Crossover, Bioequivalence Study Comparing Phase 2b 1 Mg And 5 Mg Tablet Formulations Of Cp-690,550 Under Fasted Conditions
Brief Title: A Study To Compare The Amount Of CP-690,550 That Is Absorbed Into The Blood Of Healthy Subjects Following Oral Administration Of Two Different Strength Tablets Of CP-690,550
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A3921135
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Arthritis, Rheumatoid
Keywords: Bioequivalence; healthy volunteer study; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental)
  Interventions: Drug: Treatment A; Drug: Treatment B
- Sequence 2 (Experimental)
  Interventions: Drug: Treatment B; Drug: Treatment A

INTERVENTIONS:
Drug: Treatment A — Single oral dose of 5 mg CP-690,550 administered as five 1 mg tablets (Phase 2B tablets)
  Arms: Sequence 1
Drug: Treatment B — Single oral dose of 5 mg CP-690,550 administered as one 5 mg tablet (Phase 2B tablet)
  Arms: Sequence 1
Drug: Treatment B — Single oral dose of 5 mg CP-690,550 administered as one 5 mg tablet (Phase 2B tablet)
  Arms: Sequence 2
Drug: Treatment A — Single oral dose of 5 mg CP-690,550 administered as five 1 mg tablets (Phase 2B tablets)
  Arms: Sequence 2

SUMMARY:
In this study, a 5 mg dose of CP-690,550 will be given to study subjects on two separate occasions using one of two different strength tablets each time. The amount of CP-690,550 available in the blood following administration of each tablet will be measured and compared. The overall aim of the study is to establish that a similar amount of CP-690,550 is absorbed into the blood following administration of the same dose of each different strength tablet .

DETAILED DESCRIPTION:
This is a bioequivalence study for CP-690,550.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (non-childbearing potential) subjects between the ages of 21 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >45 kg (99 lbs).
* No evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB).

Exclusion Criteria:

Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

Personal or family history of hereditary immunodeficiency (eg, severe - Evidence of any clinically significant illness, medical condition, or disease.

* Evidence or history of any clinically significant infections within the past 3 months.
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
PK parameters: AUCinf, AUClast and Cmax of CP-690,550 | PK blood samples out to 24 hours post dose in each period

SECONDARY OUTCOMES:
PK parameters: Tmax, AUCt and half-life of CP-690,550 | Derived from PK blood samples out to 24 hours post dose in each period
Safety: laboratory tests | Pre-dose on Day 0 for Period 1 and at 24 hours post last dose in each period
Safety: vital signs | Prior to dosing in each period and at 24 hours post last dose in Period 2
Safety: adverse event reporting | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921135&StudyName=A%20Study%20To%20Compare%20The%20Amount%20Of%20CP-690%2C550%20That%20Is%20Absorbed%20Into%20The%20Blood%20Of%20Healthy%20Subjects%20Following%20Oral%20Administration%20Of%20T